CLINICAL TRIAL: NCT04254224
Title: Scandinavian Diverticulitis Trial SCANDIV II: Treatment of Acute Complicated Diverticulitis: a Prospective Observational Study
Brief Title: Scandinavian Diverticulitis Trial SCANDIV-II
Acronym: SCANDIV-II
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Collaborators: Centrallasarettet Västerås (Other); Mora Hospital, Landstinget Dalarna (Unknown); Uppsala University Hospital (Other); University Hospital, Linkoeping (Other); Danderyd Hospital (Other); Sahlgrenska University Hospital (Other); Stockholm South General Hospital (Other)
Responsible Party: Principal Investigator, achabok, Ass. prof. Abbas Chabok Head of colorectal unit Surgical department Västmanlands Hospital and Centre for clinical research Uppsala University, Uppsala University
Other Study IDs: 2017/448
Record Dates: First submitted 2019-09-20; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Diverticulitis Colon
Keywords: Diverticulitis; Surgery; Hinchey; Treatment; Quality of Life
MeSH Terms: conditions — Diverticulitis, Colonic; Diverticulitis | interventions — Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diverticulitis Hinchey I-IV: Patients with complicated diverticulitis (Hinchey I-IV) treated conservatively (iv antibiotics with or without percutaneous, transrectal or transvaginal drainage) or surgically.
  Interventions: Procedure: colon resection, stoma

INTERVENTIONS:
Procedure: colon resection, stoma — oral or intravenous antibiotics treatment with or without percutanous or transrectal or transvaginal drainage
  Other Names: Conservative treatment

SUMMARY:
This study focuses on the treatment for complicated diverticulitis classified as Hinchey I-IV.

The aim of this prospective observational study is to evaluate type of treatment and the success rate of treatment in acute complicated diverticulitis (ACD) at participating hospitals in Sweden and Norway. Furthermore, the effects on quality of life for this patient group will be evaluated.

DETAILED DESCRIPTION:
Diverticular disease is among the five most common gastrointestinal disorders. Among individuals with diverticulosis the lifetime risk of suffering from diverticulitis is between 4 and 25%. The most common complications of diverticulitis are perforation, abscess formation, fistula and obstruction. Emergency surgery is necessary in up to 25% of diverticulitis patients.

The American Society of Colon and Rectal Surgeon (ASCRS, 2014) recommends abscess drainage and antibiotic treatment and later elective surgery as treatment for complicated diverticulitis, Hinchey I and II (*) for abscesses larger or equal to 5 cm while others recommend resection surgery only for Hinchey II patients. The recommendations for surgery are motivated by the belief that surgical treatment will reduce the risk for relapsing disease with intra-abdominal/pelvic sepsis by more than 40%. However, these recommendations are based on small and out-dated retrospective studies.

Perforated diverticulitis with radiologically confirmed free intraperitoneal air is a life threatening disease with significant mortality and morbidity therefore several guidelines recommend acute surgical intervention. However, a conservative non-surgical approach for the treatment of perforated diverticulitis has been shown to be effective for hemodynamically stable patients with radiologically confirmed free air. A Swedish study recently showed the incidence of complicated diverticulitis to be 9/100.000 inhabitants/year of which about one third required acute surgical intervention. The most common operation in perforated diverticulitis is Hartman's procedure, which involves removal of the involved sigmoid segment, a terminal colostomy and blind closure of the rectal stump. Also primary resection of the sigmoid colon with anastomosis is frequently used, sometimes combined with a loop-ileostomy. Laparoscopic lavage without resection has emerged as an alternative operation method. However, the SCANDIV trial showed limitations of laparoscopic lavage with a higher frequency of re-operation in the lavage group compared to primary resection after 90 days. Nevertheless, several meta-analysis based on three randomized studies showed comparable rates regarding overall mortality and morbidity in laparoscopic lavage versus resection in perforated diverticulitis.

For patients with diverticulitis complicated by fistula (colovesical, colovaginal or colo cutaneous) surgery is the recommended treatment. This condition, however, rarely presents in an acute setting.

In Scandinavia a conservative approach restricted to antibiotics and percutaneous drainage is widely accepted as solitary treatment for patients with diverticular abscesses (Hinchey I and II). Also hemodynamically stable and non-immunocompromised patients with perforated diverticulitis (Hinchey III) are often managed conservatively with antibiotics and, if required, percutaneous drainage. Acute surgical intervention is performed if the condition of the patient deteriorates during hospital stay or if the CT shows signs of faecal peritonitis (Hinchey IV). Elective surgery for patients after an episode of acute complicated diverticulitis (Hinchey I-III) is usually reserved for patients with frequent relapses or with a persisting diverticular abscess.

However, some patients have frequent relapses with abscesses which are difficult to treat and suffer for a long time until the problem is solved. This clinical experience raises the question whether the Scandinavian treatment policy might be too conservative sometimes. Although elective surgery itself can lead to new complications and eventual deterioration in quality of life, early resection might be a better option for some patients. Also the quality of life for patients after conservative management of complicated diverticulitis has not been examined in detail previously.

* I Pericolic abscess II Distant/pelvic abscess III Generalized purulent peritonitis IV Faecal peritonitis

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Clinical symptoms and laboratory results suspicious for diverticulitis
* CT findings of complicated diverticulitis with extraluminal air, presence of abscess with or without fistula or operative findings of complicated diverticulitis in an emergency setting

Exclusion Criteria:

* patients with uncomplicated diverticulitis
* unable to give informed consent.
* language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients 18 years and older with complicated diverticulitis that are admitted to hospital. Diagnosis verified with computed tomography.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-04-10 (Actual); Primary Completion 2022-04-10 (Estimated); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
Treatment in complicated diverticulitis | 1year
  Surgery or conservative managment
Treatment failure | 1year
  Complications, reoperation, readmission, recurrence , mortality

SECONDARY OUTCOMES:
Evaluation of guality of Life | 1 years
  Quality of Life according to Short Health Scale Likert-scale.
Evaluation of guality of Life | 1 years
  Quality of Life according to GIQLI.
Evaluation of guality of Life | 1 years
  Quality of Life according to EQ5D.
Stoma | 1 year
  Proportion of patients with Stoma

CONTACTS AND LOCATIONS:
Overall Officials: Abbas Chabok, MD, PhD, Principal Investigator — Uppsala University
Locations (1):
- Region Vastmanland Hospital, Västerås, Västmanland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Etzioni DA, Mack TM, Beart RW Jr, Kaiser AM. Diverticulitis in the United States: 1998-2005: changing patterns of disease and treatment. Ann Surg. 2009 Feb;249(2):210-7. doi: 10.1097/SLA.0b013e3181952888. PMID 19212172
- [Background] Sandler RS, Everhart JE, Donowitz M, Adams E, Cronin K, Goodman C, Gemmen E, Shah S, Avdic A, Rubin R. The burden of selected digestive diseases in the United States. Gastroenterology. 2002 May;122(5):1500-11. doi: 10.1053/gast.2002.32978. PMID 11984534
- [Background] Heise CP. Epidemiology and pathogenesis of diverticular disease. J Gastrointest Surg. 2008 Aug;12(8):1309-11. doi: 10.1007/s11605-008-0492-0. Epub 2008 Feb 16. PMID 18278535
- [Background] Shahedi K, Fuller G, Bolus R, Cohen E, Vu M, Shah R, Agarwal N, Kaneshiro M, Atia M, Sheen V, Kurzbard N, van Oijen MG, Yen L, Hodgkins P, Erder MH, Spiegel B. Long-term risk of acute diverticulitis among patients with incidental diverticulosis found during colonoscopy. Clin Gastroenterol Hepatol. 2013 Dec;11(12):1609-13. doi: 10.1016/j.cgh.2013.06.020. Epub 2013 Jul 12. PMID 23856358
- [Background] Morris AM, Regenbogen SE, Hardiman KM, Hendren S. Sigmoid diverticulitis: a systematic review. JAMA. 2014 Jan 15;311(3):287-97. doi: 10.1001/jama.2013.282025. PMID 24430321
- [Background] Abbas S. Resection and primary anastomosis in acute complicated diverticulitis, a systematic review of the literature. Int J Colorectal Dis. 2007 Apr;22(4):351-7. doi: 10.1007/s00384-005-0059-4. Epub 2006 Jan 7. PMID 16437211
- [Background] Feingold D, Steele SR, Lee S, Kaiser A, Boushey R, Buie WD, Rafferty JF. Practice parameters for the treatment of sigmoid diverticulitis. Dis Colon Rectum. 2014 Mar;57(3):284-94. doi: 10.1097/DCR.0000000000000075. No abstract available. PMID 24509449
- [Background] Hinchey EJ, Schaal PG, Richards GK. Treatment of perforated diverticular disease of the colon. Adv Surg. 1978;12:85-109. PMID 735943
- [Background] Ambrosetti P, Becker C, Terrier F. Colonic diverticulitis: impact of imaging on surgical management -- a prospective study of 542 patients. Eur Radiol. 2002 May;12(5):1145-9. doi: 10.1007/s00330-001-1143-y. Epub 2001 Nov 8. PMID 11976860
- [Background] Kaiser AM, Jiang JK, Lake JP, Ault G, Artinyan A, Gonzalez-Ruiz C, Essani R, Beart RW Jr. The management of complicated diverticulitis and the role of computed tomography. Am J Gastroenterol. 2005 Apr;100(4):910-7. doi: 10.1111/j.1572-0241.2005.41154.x. PMID 15784040
- [Background] Angenete E, Bock D, Rosenberg J, Haglind E. Laparoscopic lavage is superior to colon resection for perforated purulent diverticulitis-a meta-analysis. Int J Colorectal Dis. 2017 Feb;32(2):163-169. doi: 10.1007/s00384-016-2636-0. Epub 2016 Aug 27. PMID 27567926
- [Background] Ceresoli M, Coccolini F, Montori G, Catena F, Sartelli M, Ansaloni L. Laparoscopic lavage versus resection in perforated diverticulitis with purulent peritonitis: a meta-analysis of randomized controlled trials. World J Emerg Surg. 2016 Aug 30;11(1):42. doi: 10.1186/s13017-016-0103-4. eCollection 2016. PMID 27582782
- [Background] Cirocchi R, Di Saverio S, Weber DG, Tabola R, Abraha I, Randolph J, Arezzo A, Binda GA. Laparoscopic lavage versus surgical resection for acute diverticulitis with generalised peritonitis: a systematic review and meta-analysis. Tech Coloproctol. 2017 Feb;21(2):93-110. doi: 10.1007/s10151-017-1585-0. Epub 2017 Feb 15. PMID 28197792
- [Background] Marshall JR, Buchwald PL, Gandhi J, Schultz JK, Hider PN, Frizelle FA, Eglinton TW. Laparoscopic Lavage in the Management of Hinchey Grade III Diverticulitis: A Systematic Review. Ann Surg. 2017 Apr;265(4):670-676. doi: 10.1097/SLA.0000000000002005. PMID 27631772
- [Background] Elliott PA, McLemore EC, Abbass MA, Abbas MA. Robotic versus laparoscopic resection for sigmoid diverticulitis with fistula. J Robot Surg. 2015 Jun;9(2):137-42. doi: 10.1007/s11701-015-0503-6. Epub 2015 Feb 26. PMID 26531114
- [Background] Woods RJ, Lavery IC, Fazio VW, Jagelman DG, Weakley FL. Internal fistulas in diverticular disease. Dis Colon Rectum. 1988 Aug;31(8):591-6. doi: 10.1007/BF02556792. PMID 3402284
- [Background] Thorisson A, Nikberg M, Andreasson K, Smedh K, Chabok A. Non-operative management of perforated diverticulitis with extraluminal or free air - a retrospective single center cohort study. Scand J Gastroenterol. 2018 Oct-Nov;53(10-11):1298-1303. doi: 10.1080/00365521.2018.1520291. Epub 2018 Oct 24. PMID 30353758